CLINICAL TRIAL: NCT03518801
Title: Cannabidiol as an Adjunctive to Prolonged Exposure for the Treatment of PTSD
Brief Title: Cannabidiol and Prolonged Exposure
Acronym: CBD-PE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBB-001-17F
Record Dates: First submitted 2018-04-16; First posted 2018-05-08 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: PTSD
Keywords: cannabidiol; CBD; PTSD; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to one of two treatment conditions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind study. Only pharmacist will have access to randomization table.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prolonged Exposure + Cannabidiol (Experimental): Psychotherapy plus active medication
  Interventions: Behavioral: Prolonged Exposure; Drug: Cannabidiol
- Prolonged Exposure + Placebo (Active Comparator): Psychotherapy plus placebo medication
  Interventions: Behavioral: Prolonged Exposure; Drug: placebo

INTERVENTIONS:
Behavioral: Prolonged Exposure — psychotherapy
  Other Names: PE
Drug: Cannabidiol — active medication
  Other Names: CBD
  Arms: Prolonged Exposure + Cannabidiol
Drug: placebo — non-active medication
  Arms: Prolonged Exposure + Placebo

SUMMARY:
The trial will include a randomized control trial to evaluate the efficacy of using Cannabidiol (CBD), a non-intoxicating cannabinoid, as an adjunctive to Prolonged Exposure therapy (PE). The trial will compare PE + CBD to PE + placebo in a sample of 136 military Veterans with PTSD at the VA San Diego Medical Center. The study represents the logical and innovative next step for augmenting existing treatments and developing novel pharmacotherapy for PTSD. Findings from the proposed RCT will inform clinical practice and policy by investigating whether administration of CBD in the context of PE therapy will improve treatment outcomes for military Veterans with PTSD.

DETAILED DESCRIPTION:
Prolonged exposure therapy (PE) is among the most efficacious treatments for PTSD and is designated as a VA/DoD frontline treatment. However, PE does not always lead to clinically meaningful symptom reductions in Veterans with PTSD. Successful PE treatment relies on extinction learning, which is often impaired in patients with PTSD. Cannabidiol (CBD) is a non-intoxicating phytocannabinoid. Administration of specific phytocannabinoids, like CBD, increase extinction learning in patients with PTSD, and could increase the speed and effectiveness of PE therapy. CBD also modulates 5-HT1A, which may directly improve hyperarousal/insomnia symptoms, and improve engagement and retention in treatment. Given these findings, adjunctive administration of CBD+PE could improve response rates to PE and reduce the number of sessions of PE needed to reach clinically meaningful change. The proposed study is designed to test the efficacy of using CBD in conjunction with PE for the treatment of PTSD in US Military Veterans. A randomized, controlled, double-blind study will compare Veterans who receive PE+CBD to PE+placebo. Participants will include 136 male and female Veterans from all service eras with PTSD. The primary hypothesis is that PE+CBD will reduce PTSD symptoms to a greater degree than PE+placebo.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 at the time of screening.
* Judged by the study physician to be in generally good health.
* Meet clinical criteria for Posttraumatic Stress Disorder (PTSD) on the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5).
* Negative urine pregnancy test.

Exclusion Criteria:

* History of significant allergic condition, significant drug-related hypersensitivity, or allergic reaction to cannabinoids.
* Used cannabis, synthetic cannabinoid, cannabinoid analogue, or any CBD or THC-containing product within 30 days of eligibility screening.
* Patient has had a change in psychopharmacotherapy regimen in the last 4 weeks, or has any plans to change regimen over the course of the study.
* Patient is engaged in trauma-related psychotherapy for PTSD.
* Current or past DSM-5 diagnosis of dissociative identity disorder, eating disorder with active purging, personality disorders, primary psychotic disorder, or bipolar affective disorder type 1.
* Patient is currently prescribed medications with possible CBD-drug interactions.
* History of actual suicide attempt in the last 5 years.
* Unmanaged obstructive sleep apnea.
* Positive drug screen for THC, barbiturates, amphetamines (if not prescribed), benzodiazepines, and/or opiates.
* History of treatment for, or evidence of, moderate to severe alcohol or drug abuse within the past year or regular alcohol consumption exceeding recommended limits.
* Lifetime history of Cannabis Use Disorder.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale DSM 5 (CAPS-5) | Baseline, Post Treatment (16-weeks), 1-Month Follow-up (20-weeks), 3-Month Follow-up (28-weeks)
  Change in PTSD Symptoms will be assessed by change in Total Severity Score (summed severity ratings on items 1-20) on the Clinician-Administered PTSD Scale DSM 5 (CAPS-5); CAPS-5 Total Severity scores range from 0 to 80; Higher scores indicate higher severity.

SECONDARY OUTCOMES:
PTSD Checklist (PCL-5) | Baseline, Weekly (up to 16-weeks)
  Rate of PTSD symptom reduction will be assessed by comparing the time-to-event of clinical response to treatment. The time-to-event is defined by number of PE sessions completed before patient achieves a 10-point reduction from baseline in total (summed) PTSD Checklist scores (PCL-5). PCL-5 Total Scores range from 0 to 80; Higher scores indicate worse functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine R Ayers, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA; Brian Martis, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No